CLINICAL TRIAL: NCT06407791
Title: Clinical Evaluation of a Device for Treatment of Lymphedema of the Upper Extremity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-22-1780
Record Dates: First submitted 2024-04-08; First posted 2024-05-09 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- LymphaVibe Experimental Arm (Experimental): All patients in this single arm (only arm of the study) will receive both treatment with the LymphaVibe AND the standard of care, thus serving as their own control. Patients will have baseline measurements taken, receive treatment with the LymphaVibe, have their measurements repeated, receive the standard of care, and have their measurements repeated again.
  Interventions: Device: LymphaVibe

INTERVENTIONS:
Device: LymphaVibe — The LymphaVibe is a newly-developed device that uses a vibratory sequence to gently move stagnant lymphatic fluid from the arm to the nearest group of functioning lymph nodes

SUMMARY:
Lymphedema is a painful and disfiguring condition related to the buildup of protein-rich fluid in the body's tissues. The goal of this research study is to determine the safety and efficacy of a novel, proprietary device in the treatment of upper extremity lymphedema. This device has been previously studied on healthy people that do not have a diagnosis of lymphedema. It was found that using the device on them does not cause significant changes to their vital signs or level of pain. Side effects are reported sometimes; however, these are to be expected and are also frequently reported when people receive the standard of care for their lymphedema. Patients who have diagnosed lymphedema will be approached to participate in this study as part of their care. Participants will wear this device for approximately 40 minutes and then have certain measurements taken before and after doing so. These measurements include the size of their arm, how much pain/discomfort they are currently in, and if they experienced any side effects. After getting treatment with the device, they will receive the standard of care treatment for their lymphedema from their provider. After the standard of care has concluded, the previously mentioned measurements will be repeated. This data will be put together and analyzed to look for differences in arm size before and after treatment with the device as well as to look for the prevalence of side effects.

DETAILED DESCRIPTION:
For each study visit, participants will be asked to arrive 45 minutes before the beginning of their regularly scheduled follow-up visit. Research activities will take 45 minutes.

Upon early arrival to their regularly scheduled appointment, participants will be fitted for their very own, "athletic sleeve" by a member of the research team. This athletic sleeve will be used throughout the duration of the study. Participants will be asked to come wearing a tank top or short-sleeved t-shirt. If they do not come dressed as such, they will have the opportunity to change in a private space.

Before donning the athletic sleeve, a member of the research team will measure the participant's upper limb circumference and induration and administer a baseline survey using the first section of the Lymphedema Life Impact Scale (LLIS - document attached). Upper extremity circumference will be measured in centimeters at several points, which are: palmar crease, the wrist below the styloid process, wrist + 10 cm, wrist + 20 cm, wrist + 30 cm, and wrist + 40 cm. Upper extremity induration will be measured at the same points as circumference. These measurements are being taken solely for research purposes and should take approximately 3 minutes.

The athletic sleeve will be donned by the participant and the novel therapeutic device will be placed over it. A standardized sequence of vibratory therapy will be applied. Use of this device will not impact standard of care in any way. The participant may ask to stop the research session at any time

The athletic sleeve will then be removed, and a member of the research team will measure the participant's upper limb circumference and induration and administer a survey using the first section of the Lymphedema Life Impact Scale. These measurements are being taken solely for research purposes and should take approximately 3 minutes. Participants will be asked if they experienced any side effects or adverse effects.

Standardized decongestive therapy will be performed by qualified personnel. This step takes approximately 1 hour and would happen regardless or whether or not patients are enrolled in this study. At the conclusion of the standardized decongestive therapy, the measurements and surveys mentioned previously will be repeated. Participants will also be asked if they experienced any side effects with the standard of care treatment.

This series of steps will be repeated at the participants' weekly follow-up visits for four weeks. Standardized decongestive therapy for lymphedema is most often performed on a weekly basis (and is one of the inclusion criteria for this study). Therefore, choosing this visit frequency would not greatly alter a participant's schedule or ability to perform other daily tasks.

If a participant chooses to withdraw from the study early or needs to be removed from the study for their own safety, notes will be added to research documentation and the patient's electronic medical chart indicating their departure from the study. Going forward, they would receive standard decongestive therapy as before their participation in the study.

Study subject limb circumference, induration data, and survey data will be analyzed using a paired t-test.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Clinical diagnosis of lymphedema
* Receiving current, once weekly, lymphedema treatment by Physical Therapist(PT)/Occupational Therapist (OT)
* Participants must have the ability to provide consent for themselves

Exclusion Criteria:

* Active infection
* Active cancer (not in remission)
* Diagnosis of/past medical history of Deep Vein Thrombosis (DVT) or Pulmonary Embolism (PE)
* Active phlebitis
* Diagnosis of Congestive Heart Failure (CHF)
* Previous severe trauma (i.e. requiring extensive corrective surgery)
* History of vascular surgery
* Lesions of the skin or weeping in the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Rates of reported side effects | Weekly for 4 weeks
  Will be assessed by recording rates of side effects reported by study subjects
Device efficacy in reducing lymphedema burden | Weekly for 4 weeks
  Will be assessed by recording changes in upper extremity circumference (cm)
Device efficacy in reducing lymphedema burden | Weekly for 4 weeks
  Will be assessed by recording changes in upper extremity induration
Device efficacy in reducing lymphedema burden | Weekly for 4 weeks
  Will be assessed by recording changes in the first section of the Lymphedema Life Impact Scale (LLIS) score that deals with physical symptoms of lymphedema only

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Brown, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Clinic, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nimmana BK, Kimyaghalam A, Manna B. Lymphedema. 2025 Oct 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537239/ PMID 30725924

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06407791/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT06407791/ICF_001.pdf